## The role of Ovarian PRP Therapy in Poseidon Poor Responders Women undergoing ICSI Cycle

University of Kerbala College of Medicine Medical Research Bioethical Committee

No: 25 - 8

Date: 12/1/2025



APPROVAL LETTER

Itlal Jummha Abudl Rasool Al Asadi Imam Al Hassan Teaching Hospital, Karbala Health Directorate

Title of Project: "The impact of ovarian PRP in Poseidon poor responders women undergoing ICSI cycle"

This is to certify that proposal provided have satisfactorily addressed the research bioethical guidelines.

Please consider the following requirements of approval:

- 1. Approval will be valid for one year. By the end of this period, if the project has been completed, abandoned, altered, discontinued or not commenced for any reason, you are required to announce to the Committee. And you should inform the committee if the study extends over one year.
- 2. You must notify the Committee immediately in the event of any adverse effects on participants or of any unforeseen events that might affect continued ethical acceptability of the project.
- 3. All participants must be informed about the research issue and objective, taking their consent to participate. Always consider the confidentiality of personal information and/or opinions, and they must never be obligated to participate and explaining the value and benefits of their participation.
- 4. At all times you are responsible for the ethical conduct of your research in accordance with the standard bioethical guidelines. In agreement with WMA Declaration of Helsinki - Ethical Principles for Medical Research Involving Human Participants.
- 5. The Committee should be notified if you will be applying for or have applied for internal or external funding for the above project.
- 6. All participants must be informed about the research issue and objectives prior to intervention or taking blood samples which should be voluntary and no extra costs charged on them.
- 7. This document does not compensate administrative or ethical approval might be required from Karbala Health Directorate, Hospitals or other bodies.

Ali Slife Professor Dr. Ali A. Abutiheen

Chair, Medical Research Bioethical Committee

College of Medicine - University of Kerbala